CLINICAL TRIAL: NCT06579612
Title: The Benefits of Individualized Follow-up With a Sport-Health Professional in the Care of Patients With Chronic Respiratory Diseases, to Maintain Long-term Benefits After a Respiratory Rehabilitation Program
Brief Title: The Benefits of Individualized Follow-up With a Sport-Health Professional in the Care of Patients With Chronic Respiratory Diseases
Acronym: WANTTOMOVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 29BRC22.0256
Record Dates: First submitted 2024-08-26; First posted 2024-08-30 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Chronic Respiratory Disease
Keywords: chronic respiratory disease; pulmonary rehabilitation
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Randomized controlled superiority trial in parallel arms (1:1 ratio) comparing personalized follow-up and support after a pulmonary rehabilitation program (experimental group) versus a control group receiving only usual care,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (No Intervention): Patient in the control arm will beneficiate from commun practice
- Experimental arm (Experimental): Patient in the control arm will beneficiate from a personalized follow-up and support after a pulmonary rehabilitation program
  Interventions: Other: Personalized follow-up and support

INTERVENTIONS:
Other: Personalized follow-up and support — After a pulmonary rehabilitation program, an interview with a professional will enable the professional to identify the barriersand enablers of physical activity engagement, and to identify (with the patient) a plan for maintaining a physical activities adapted in daily life. Adapted solutions will then be proposed.
  Arms: Experimental arm

SUMMARY:
Pulmonary rehabilitation is an integral part of care for patients with chronic respiratory diseases. It improves patients' physical capacities, quality of life and symptoms, at least in the short term.

The hypothesis that patients receiving personalized support from a professional following pulmonary rehabilitation will maintain long-term benefits.

This study concerns patients with a diagnosis of one or more chronic respiratory diseases.

It is a multicenter, blinded, randomized controlled superiority trial in 2 parallel arms:

* a group comparing follow-up and personalized support after a pulmonary rehabilitation program (experimental group)
* a control group receiving only usual care

DETAILED DESCRIPTION:
Pulmonary rehabilitation is an integral part of care for patients with chronic respiratory diseases. It improves patients' physical capacities, quality of life and symptoms, at least in the short term.

The hypothesis that patients receiving personalized support from a professional following pulmonary rehabilitation will maintain long-term benefits.

This study concerns patients with a diagnosis of one or more chronic respiratory diseases.

It is a multicenter, blinded, randomized controlled superiority trial in 2 parallel arms:

* a group comparing follow-up and personalized support after a pulmonary rehabilitation program (experimental group)
* a control group receiving only usual care

Each patient is followed up for 24 months with a visit every 6 months. A total of 352 subjects will be recruited

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one or more chronic respiratory diseases (asthma, chronic obstructive pulmonary disease, diffuse interstitial lung disease, bronchiectasis, obstructive sleep apnea syndrome, etc.).
* Participation in a respiratory pulmonary program
* Have given consent
* Patient of legal age
* Patient affiliated to Social Security

Exclusion Criteria:

* Any medical contraindication to the practice of adapted physical activity in rehabilitation
* Patients under guardianship or curatorship
* Patients deprived of their liberty
* Patients over 80 years of age at the time of inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2029-11-07 (Estimated); Study Completion 2029-11-07 (Estimated)

PRIMARY OUTCOMES:
Difference in average number of daily steps | At inclusion (V1) and at 24 Months (V5)
  The difference in average daily steps measured by accelerometry (over 7 days) at the end of the pulmonary rehabilitation course (V1) and after 24 months of personalized follow-up (V5).

SECONDARY OUTCOMES:
Cost-utility comparison between the two groups | At 24 Months (V5)
  The cost-utility comparison between the two groups at 24 months was carried out by means of a medico-economic evaluation. This evaluation contains 5 items : direct medical costs; costs of care in the experimental group; incremental cost-utility ratio at 24 months; medical indicator results measured in QALYs and health-related quality of life.
Comparison of changes in physical activity levels between the two groups | At 24 Months (V5)
  the evolution of physical activity levels is assessed with levels of activity :
  * Sedentary time (min/day)
  * Time spent in activity with light intensity (min/day)
  * Time spent in activity with moderate intensity (min/day)
  * Time spent in activity with vigorous intensity (min/day)
Comparison of changes in physical capacities between the two groups | A 24 Months (V5)
  The evolution of physical capacities is assessed with walking distance measured in the 6-minute walk test.
  The 6-minute walk test: total walked distance (in metres). The test will be performed twice, the best performance will be kept as reference value.
Comparison of changes in physical capacities between the two groups | A 24 Months (V5)
  The evolution of physical capacities is assessed with the endurance time on ergocycle at 80% of peak power, in seconds.
Comparison of changes in physical capacities between the two groups | A 24 Months (V5)
  The evolution of physical capacities is assessed with the quadriceps strength measured in the maximal isometric contraction test.
Comparison of changes in symptoms between the two groups | At 24 Months (V5)
  The evolution of symptoms is assessed with dyspnoea score (DYSPNEA-12). The DYSPNEA-12 comprised of 12 different breathlessness descriptors with each scored on a four-item scale (none-0, mild-1, moderate2, severe-3). Item scores are summed (D-12 Total) and can be divided into sub-scores reflecting Physical and Affective domains.
Comparison of changes in psychological dimensions between the two groups | At 24 Months (V5)
  The evolution of psychological dimensions is assessed with the motivation scores according to different levels of regulation assessed by the Motivation for Physical Activity for Health Purposes Scale (EMAPS). This questionnaire includes 18 items. The EMAPS is used to evaluate the motivation to practice physical activities. The answer to questions goes from 1 to 7 with 1 (does not match at all) and 7 (matches very strongly).
Comparison of changes in psychological dimensions between the two groups | At 24 Months (V5)
  The evolution of psychological dimensions is assessed with the anxiety and depression scores using the Hospital Anxiety and Depression scale (HAD). This questionnaire includes 7 items for depression and 7 items for anxiety. Each item had been answered by the patient on a four point (0-3) response category so the possible scores ranged from 0 to 21 for anxiety and for depression. A score of 0 to 7 for either subscale could be regarded as being in the normal range, a score of 11 or higher indicating probable presence ('caseness') of the mood disorder and a score of 8 to 10 being just suggestive of the presence of the respective state.
Comparison of changes in health indicator between the two groups | At 24 Months (V5)
  The evolution of health indicator is assessed with a St George's Respiratory Questionnaire (SGRQ). This questionnaire comprises 3 components: the symptom component assesses the effects of respiratory symptoms, their frequency and severity, the activity component looks at activities that cause and/or are limited by breathlessness, and the impact component assesses the disruption to social and psychological functioning induced by the disease. The total score ranges from 100 (low quality of life) to 0 (excellent quality of life).
Comparison of changes in quality of life indicator between the two groups | At 24 Months (V5)
  The evolution of quality of life indicator is assessed with EuroQol " five dimensions questionnaire " (EQ5DL). EQ5DL is a questionnaire including 5 items mobility, personal care, usual activities, pain/discomfort and anxiety/depression.
Comparison of changes in parameters (barriers and levers to physical activity) between the two groups | At 24 Months (V5)
  The evolution of parameters (barriers and levers to physical activity) is assessed with the socioeconomic investigation results. This questionnaire was created for this study to gather information on the socio-economic and environmental profile of people in relation to the practice of physical activity (Barriers and levers to practice, transportation, cost of practicing physical activity, place of practice).
Comparison of changes in physical capacities between the two groups | At 24 Months (V5)
  The evolution of physical capacities is assessed with the Forced Expiratory Volume in 1 Second measured by spirometry
Comparison of changes in physical capacities between the two groups | At 24 Months (V5)
  The evolution of physical capacities is assessed with the Forced Vital Capacity measured by spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Agnès GIROUX-METGES, MD, PhD, Principal Investigator — Brest Universty Hospital
Locations (2):
- France (2):
  - CHU de Brest, Brest
  - CH des Pays de Morlaix, Morlaix

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement